CLINICAL TRIAL: NCT03950674
Title: A Randomized, Double-Blind, Phase III Study of Platinum+Pemetrexed Chemotherapy With or Without Pembrolizumab (MK-3475) in First Line Metastatic Non-squamous Non-small Cell Lung Cancer Subjects (KEYNOTE-189)
Brief Title: Study of Pemetrexed+Platinum Chemotherapy With or Without Pembrolizumab (MK-3475) in Participants With First Line Metastatic Nonsquamous Non-small Cell Lung Cancer (MK-3475-189/KEYNOTE-189)-Japan Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3475-189 Japan Extension; 163421 (Registry Identifier: JAPIC-CTI); MK-3475-189 (Other: Merck); KEYNOTE-189 (Other: Merck)
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-05

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Non-Small-Cell Lung Cancer (NSCLC); PD1; PD-1; PDL1; PD-L1; Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Cisplatin; Carboplatin; Pemetrexed; Folic Acid; Vitamin B 12; Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab with Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) PLUS pemetrexed 500 mg/m^2 IV (with vitamin supplementation) PLUS cisplatin 75 mg/m^2 IV OR carboplatin Area Under the Curve (AUC) 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by pembrolizumab 200 mg IV PLUS pemetrexed 500 mg/m^2 IV Q3W until progression. Participants who receive pembrolizumab 200 mg IV Q3W for up to 2 years, but experience disease progression, are eligible to receive a second course of pembrolizumab monotherapy 200 mg IV Q3W, at the investigator's discretion, for up to another year.
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Dietary Supplement: Folic acid 350-1000 μg; Dietary Supplement: Vitamin B12 1000 μg; Drug: Dexamethasone 4 mg
- Placebo with Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed (Active Comparator): Participants receive saline placebo IV PLUS pemetrexed 500 mg/m^2 IV (with vitamin supplementation) PLUS cisplatin 75 mg/m^2 IV OR carboplatin AUC 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by saline placebo IV PLUS pemetrexed 500 mg/m^2 IV Q3W until progression. Participants who receive saline placebo, but experience disease progression, can switch over to pembrolizumab monotherapy 200 mg IV Q3W, at the investigator's discretion, for up to 2 years. The participants who switch over to pembrolizumab 200 mg IV Q3W, but experience disease progression, are eligible to receive a second course of pembrolizumab monotherapy 200 mg IV Q3W, at the investigator's discretion, for up to another year.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Dietary Supplement: Folic acid 350-1000 μg; Dietary Supplement: Vitamin B12 1000 μg; Drug: Dexamethasone 4 mg; Drug: Saline solution

INTERVENTIONS:
Biological: Pembrolizumab 200 mg — IV infusion
  Arms: Pembrolizumab with Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed
Drug: Cisplatin — IV infusion
Drug: Carboplatin — IV infusion
Drug: Pemetrexed — IV infusion
Dietary Supplement: Folic acid 350-1000 μg — Orally; at least 5 doses of folic acid must be taken during the 7 days preceding the first dose of pemetrexed, and folic acid dosing must continue during the full course of therapy and for 21 days after the last dose of pemetrexed.
Dietary Supplement: Vitamin B12 1000 μg — Intramuscular injection in the week preceding the first dose of pemetrexed and once every 3 cycles thereafter. Subsequent vitamin B12 injections may be given the same day as pemetrexed administration.
Drug: Dexamethasone 4 mg — For prophylaxis; orally twice per day (or equivalent). Taken the day before, day of, and day after pemetrexed administration.
Drug: Saline solution — IV infusion
  Arms: Placebo with Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed

SUMMARY:
This is a Japan Extension Study of Global Study MK-3475-189 (NCT02578680). This is an efficacy and safety study of pembrolizumab (MK-3475) combined with pemetrexed/platinum chemotherapy versus pemetrexed/platinum chemotherapy alone in adult Japanese participants with advanced or metastatic nonsquamous non-small cell lung cancer (NSCLC) who have not previously received systemic therapy for advanced disease. Participants will be randomly assigned to receive pembrolizumab combined with pemetrexed/platinum (Investigators choice of cisplatin or carboplatin), OR pemetrexed/platinum (Investigators choice of cisplatin or carboplatin).

With Amendment 11 (effective date 31-Jan-2022), once the study objectives have been met or the study has ended, participants will be discontinued from this study and will be enrolled in an extension study to continue protocol-defined assessments and treatment.

The primary hypothesis is that pembrolizumab in combination with pemetrexed/platinum chemotherapy prolongs Progression-Free Survival (PFS) and Overall Survival (OS) compared to pemetrexed/platinum chemotherapy alone.

DETAILED DESCRIPTION:
The MK-3475-189-Japan Extension Study will be identical to the global study (e.g. inclusion and exclusion criteria, study primary and secondary outcome measures and study procedures).

The MK-3475-189-Japanese Extension Study enrolled a total of 30 participants and the analyses included 10 participants (pembrolizumab =4; control = 6) that had been previously enrolled in the MK-3475-189 global study (NCT02578680), resulting in a total of 40 participants.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically-confirmed or cytologically confirmed diagnosis of stage IV nonsquamous NSCLC.
* Has confirmation that epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK)-directed therapy is not indicated.
* Has measurable disease.
* Has not received prior systemic treatment for their advanced/metastatic NSCLC.
* Can provide tumor tissue.
* Has a life expectancy of at least 3 months.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
* Has adequate organ function
* If female of childbearing potential, is willing to use adequate contraception for the course of the study through 120 days after the last dose of study medication or through 180 days after last dose of chemotherapeutic agents.
* If male with a female partner(s) of child-bearing potential, must agree to use adequate contraception starting with the first dose of study medication through 120 days after the last dose of study medication or through 180 days after last dose of chemotherapeutic agents.

Exclusion Criteria:

* Has predominantly squamous cell histology NSCLC.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to administration of pembrolizumab.
* Before the first dose of study medication: a) Has received prior systemic cytotoxic chemotherapy for metastatic disease, b) Has received antineoplastic biological therapy (e.g. erlotinib, crizotinib, cetuximab), c) Had major surgery (<3 weeks prior to first dose)
* Received radiation therapy to the lung that is >30 Gray (Gy) within 6 months of the first dose of study medication.
* Completed palliative radiotherapy within 7 days of the first dose of study medication.
* Is expected to require any other form of antineoplastic therapy while on study.
* Received a live-virus vaccination within 30 days of planned start of study medication.
* Has clinically active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction, peritoneal carcinomatosis.
* Known history of prior malignancy except if participant has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy, except for successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Previously had a severe hypersensitivity reaction to treatment with another monoclonal antibody (mAb).
* Known sensitivity to any component of cisplatin, carboplatin or pemetrexed.
* Has active autoimmune disease that has required systemic treatment in past 2 years.
* Is on chronic systemic steroids.
* Is unable to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs), other than an aspirin dose ≤1.3 g per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam).
* Is unable or unwilling to take folic acid or vitamin B12 supplementation.
* Had prior treatment with any other anti-programmed cell death-1 (PD-1), or PD-ligand 1 (PD-L1) or PD-L2 agent or an antibody targeting other immuno-regulatory receptors or mechanisms. Has participated in any other pembrolizumab study and has been treated with pembrolizumab.
* Has an active infection requiring therapy.
* Has known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B or C.
* Has known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial.
* Is a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
* Has symptomatic ascites or pleural effusion.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2023-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (10):
- Japan (10):
  - National Hospital Organization Nagoya Medical Center ( Site 0324), Nagoya, Aichi-ken
  - Kurume University Hospital ( Site 0326), Kurume, Fukuoka
  - Hyogo Cancer Center ( Site 0325), Akashi, Hyōgo
  - Kanazawa University Hospital ( Site 0328), Kanazawa, Ishikawa-ken
  - Kansai Medical University Hospital ( Site 0313), Hirakata, Osaka
  - Shizuoka Cancer Center Hospital and Research Institute ( Site 0322), Sunto-gun, Shizuoka
  - National Hospital Organization Shikoku Cancer Center ( Site 0303), Matsuyama
  - Okayama University Hospital ( Site 0327), Okayama
  - National Cancer Center Hospital ( Site 0301), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 0323), Tokyo

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Horinouchi H, Nogami N, Saka H, Nishio M, Tokito T, Takahashi T, Kasahara K, Hattori Y, Ichihara E, Adachi N, Noguchi K, Souza F, Kurata T. Pembrolizumab plus pemetrexed-platinum for metastatic nonsquamous non-small-cell lung cancer: KEYNOTE-189 Japan Study. Cancer Sci. 2021 Aug;112(8):3255-3265. doi: 10.1111/cas.14980. Epub 2021 Jun 15. PMID 34036692
- [Derived] Cheng Y, Yang JC, Okamoto I, Zhang L, Hu J, Wang D, Hu C, Zhou J, Wu L, Cao L, Liu J, Zhang H, Sun H, Wang Z, Gao H, Yan Y, Xiao S, Lin J, Pietanza MC, Kurata T. Pembrolizumab plus chemotherapy for advanced non-small-cell lung cancer without tumor PD-L1 expression in Asia. Immunotherapy. 2023 Sep;15(13):1029-1044. doi: 10.2217/imt-2023-0043. Epub 2023 Jul 19. PMID 37465924
- [Derived] Rolfo C, Hess LM, Jen MH, Peterson P, Li X, Liu H, Lai Y, Sugihara T, Kiiskinen U, Vickers A, Summers Y. External control cohorts for the single-arm LIBRETTO-001 trial of selpercatinib in RET+ non-small-cell lung cancer. ESMO Open. 2022 Aug;7(4):100551. doi: 10.1016/j.esmoop.2022.100551. Epub 2022 Aug 2. PMID 35930972
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Japanese Extension study for MK-3475-189 enrolled a total of 30 participants and the analyses included 10 participants (pembrolizumab =4; control = 6) that had been previously enrolled in the global study for MK-3475-189 (NCT02578680), resulting in a total of 40 participants.
Pre-assignment Details: Four participants randomized to placebo treatment had switched over to receive pembrolizumab monotherapy. Participants receiving pembrolizumab in the first course and those who switched over from placebo to pembrolizumab were eligible to receive a second course of pembrolizumab if they met certain criteria. Data from the second course treatment contributed to safety data only. Final analyses for all primary and secondary outcome measures were done at the protocol-specified cutoff (20-May-2019).
Groups:
- Pembrolizumab With Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed: Participants received pembrolizumab 200 mg intravenously (IV) PLUS pemetrexed 500 mg/m^2 IV (with vitamin supplementation) PLUS cisplatin 75 mg/m^2 IV OR carboplatin Area Under the Curve (AUC) 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by pembrolizumab 200 mg IV PLUS pemetrexed 500 mg/m^2 IV Q3W until progression. Participants who received pembrolizumab 200 mg IV Q3W for up to 2 years, but experienced disease progression, were eligible to receive a second course of pembrolizumab monotherapy 200 mg IV Q3W, at the investigator's discretion, for up to another year.
- Placebo With Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed: Participants received saline placebo IV PLUS pemetrexed 500 mg/m^2 IV (with vitamin supplementation) PLUS cisplatin 75 mg/m^2 IV OR carboplatin AUC 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by saline placebo IV PLUS pemetrexed 500 mg/m^2 IV Q3W until progression. Participants who received saline placebo, but experienced disease progression, were switched over to pembrolizumab monotherapy 200 mg IV Q3W, at the investigator's discretion, for up to 2 years. The participants who had switched over to pembrolizumab 200 mg IV Q3W, but experienced disease progression, were eligible to receive a second course of pembrolizumab monotherapy 200 mg IV Q3W, at the investigator's discretion, for up to another year.
Period: Overall Study
Arm/Group | Pembrolizumab With Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed | Placebo With Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed
Started | 25 | 15
Treated | 25 | 15
Switched to Pembrolizumab Monotherapy | 0 | 4
Second Course Treatment With Pembrolizumab Monotherapy | 1 | 0
Completed | 0 | 0
Not Completed | 25 | 15
Not completed — Death | 16 | 15
Not completed — Participation in the study terminated by the sponsor | 9 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab With Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed | Placebo With Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed | Total
Number analyzed (Participants) | 25 | 15 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (12.7) | 60.9 (11.8) | 60.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 19 | 12 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 15 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 25 | 15 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Programmed Cell Death-Ligand 1 (PD-L1) Tumor Status [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from an archival or newly obtained biopsy. Participants with a TPS ≥1% were classified as PD-L1 positive and participants with a TPS <1% were classified as PD-L1 negative.
  Participants
    TPS <1% | 14 | 6 | 20
    TPS ≥1% | 10 | 6 | 16
    Not Evaluable | 1 | 3 | 4
Platinum Chemotherapy [Count of Participants; unit: Participants] — Participants were classified according to the type of platinum chemotherapy the Investigator chose for them to receive: Cisplatin or Carboplatin.
  Participants
    Cisplatin | 18 | 8 | 26
    Carboplatin | 7 | 7 | 14
Smoking Status [Count of Participants; unit: Participants] — Participants were classified according to their smoking status: Never Smoker or Former/Current Smoker.
  Participants
    Never Smoker | 7 | 3 | 10
    Former/Current Smoker | 18 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as Assessed by Blinded Central Imaging
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 is presented.
Time Frame: Up to approximately 31 months
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab With Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed | Placebo With Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed
Number analyzed (Participants) | 25 | 15
Months | 16.5 [8.8 to 21.1] | 7.1 [4.7 to 21.4]
Statistical Analysis 1: Comparison: Pembrolizumab With Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed vs Placebo With Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed; Test type: Other; p = 0.12511, Log Rank — One-sided p-value based on unstratified log-rank test; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.27 to 1.42] — Based on Cox regression model with treatment as a covariate stratified by PD-L1 status (≥1% vs. <1%), platinum chemotherapy (cisplatin vs. carboplatin) & smoking status (never vs. former/current). Pembrolizumab=numerator; Control=denominator

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up. The OS is presented.
Time Frame: Up to approximately 31 months
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab With Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed | Placebo With Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed
Number analyzed (Participants) | 25 | 15
Months | NA [NA to NA] — NA=Median OS not reached NA=Lower Limit OS not reached NA=Upper Limit OS not reached | 25.9 [11.9 to 29.0]
Statistical Analysis 1: Comparison: Pembrolizumab With Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed vs Placebo With Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed; Test type: Other; p = 0.03127, Log Rank — One-sided p-value based on unstratified log-rank test; Hazard Ratio (HR) = 0.29, 95% CI 2-sided [0.07 to 1.15] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Response Rate (ORR) Per RECIST 1.1 as Assessed by Blinded Central Imaging
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1. The percentage of participants who experienced a CR or PR is presented.
Time Frame: Up to approximately 31 months
Population: The analysis population consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab With Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed | Placebo With Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed
Number analyzed (Participants) | 25 | 15
Percentage of Participants | 56.0 [34.9 to 75.6] | 33.3 [11.8 to 61.6]

4. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Assessed by Blinded Central Imaging
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of a CR or PR until PD or death. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. DOR assessments were based on blinded central imaging review with confirmation. The DOR per RECIST 1.1 for all participants who experienced a confirmed CR or PR is presented.
Time Frame: Up to approximately 31 months
Population: The analysis population consisted of all randomized participants who experienced a confirmed CR or confirmed PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab With Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed | Placebo With Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed
Number analyzed (Participants) | 14 | 5
Months | 13.6 [5.9 to 19.6] | 9.7 [3.4 to NA] — NA=Upper Limit DOR not reached

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event was defined as any untoward medical occurrence in a clinical study participant administered a pharmaceutical product which did not necessarily have a causal relationship with this treatment. An adverse event was any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that was temporally associated with the use of the study drug was also an adverse event. Per protocol, final analysis for this outcome measure was performed for the first course of pembrolizumab or placebo treatment. The number of participants who experienced an AE is reported.
Time Frame: Up to approximately 24 months
Population: The analysis population consisted of all randomized participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab With Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed | Placebo With Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed
Number analyzed (Participants) | 25 | 15
Participants | 25 | 15

6. Secondary Outcome: Number of Participants Who Discontinued Any Study Drug Due to an AE
Description: An adverse event was defined as any untoward medical occurrence in a clinical study participant administered a pharmaceutical product which did not necessarily have a causal relationship with this treatment. An adverse event was any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that was temporally associated with the use of the study drug was also an adverse event. Per protocol, final analysis for this outcome measure was performed for the first course of pembrolizumab or placebo treatment. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 21 months
Population: The analysis population consisted of all randomized participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab With Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed | Placebo With Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed
Number analyzed (Participants) | 25 | 15
Participants | 9 | 3

7. Other Pre Specified Outcome: Progression-Free Survival (PFS) as Assessed by Investigator Immune-related RECIST (irRECIST) Response Criteria
Description: PFS was defined as the time from randomization to the first documented immune-related progressive disease (irPD) or death due to any cause, whichever occurred first. Per irRECIST, irPD was confirmed if any of the following are observed in 2 scans performed at least 4 weeks apart: target lesion sum of diameters remains ≥20 % and at least 5 mm absolute increase compared to nadir; non-target disease resulting in initial PD is qualitatively worse; new lesion resulting in initial irPD is qualitatively worse; additional new lesion(s) since last evaluation; or additional new non-target lesion progression since last evaluation. The PFS per irRECIST 1.1 is presented.
Time Frame: Up to approximately 31 months
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab With Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed | Placebo With Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed
Number analyzed (Participants) | 25 | 15
Months | 13.7 [6.4 to 22.0] | 7.6 [2.6 to 11.9]

ADVERSE EVENTS:
Time Frame: Up to approximately 80 months
Description: All participants who received ≥1 dose of treatment. Per protocol, disease progression was not considered an adverse event (AE) unless treatment related. Medical Dictionary for Regulatory Activities (MedDRA) terms neoplasm progression (NP), malignant NP, and disease progression not related to treatment were excluded. All-cause mortality and AEs analyzed for both study arms, participants switched over from placebo to pembrolizumab, and those who received second course pembrolizumab if applicable.
Groups:
- Placebo Switched Over to Pembrolizumab Monotherapy: Qualified participants who received saline placebo with pemetrexed and platinum chemotherapy followed by placebo and pemetrexed, and who experienced disease progression, were switched over to receive pembrolizumab monotherapy 200 mg IV on Day 1 Q3W for up to 2 years.
- Second Course Treatment for the Pembrolizumab With Pemetrexed and Platinum Chemotherapy Arm: Participants who received pembrolizumab with pemetrexed and platinum chemotherapy followed by pembrolizumab and pemetrexed during the initial treatment, and met certain criteria, initiated a second course of pembrolizumab monotherapy at 200 mg IV Q3W for up to 1 additional year.
- Second Course Treatment for the Placebo Switched Over to Pembrolizumab Monotherapy Arm: Participants who were switched from saline placebo to receive pembrolizumab monotherapy, and met certain criteria, initiated a second course of pembrolizumab monotherapy at 200 mg IV Q3W for up to 1 additional year.
Arm/Group | Pembrolizumab With Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed | Placebo With Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed | Placebo Switched Over to Pembrolizumab Monotherapy | Second Course Treatment for the Pembrolizumab With Pemetrexed and Platinum Chemotherapy Arm | Second Course Treatment for the Placebo Switched Over to Pembrolizumab Monotherapy Arm
All-Cause Mortality (participants affected / at risk) | 15/25 | 11/15 | 4/4 | 1/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 9/25 | 6/15 | 1/4 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 25/25 | 15/15 | 4/4 | 0/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab With Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed (N=25) | Placebo With Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed (N=15) | Placebo Switched Over to Pembrolizumab Monotherapy (N=4) | Second Course Treatment for the Pembrolizumab With Pemetrexed and Platinum Chemotherapy Arm (N=1) | Second Course Treatment for the Placebo Switched Over to Pembrolizumab Monotherapy Arm (N=0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
Pyrexia (General disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | NA
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Oesophageal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | NA
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab With Pemetrexed and Platinum Chemotherapy Followed by Pembrolizumab and Pemetrexed (N=25) | Placebo With Pemetrexed and Platinum Chemotherapy Followed by Placebo and Pemetrexed (N=15) | Placebo Switched Over to Pembrolizumab Monotherapy (N=4) | Second Course Treatment for the Pembrolizumab With Pemetrexed and Platinum Chemotherapy Arm (N=1) | Second Course Treatment for the Placebo Switched Over to Pembrolizumab Monotherapy Arm (N=0)
Anaemia (Blood and lymphatic system disorders) | 11 (17) | 10 (11) | 0 (0) | 0 (0) | NA
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 7 (13) | 0 (0) | 0 (0) | NA
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | NA
Neutropenia (Blood and lymphatic system disorders) | 3 (5) | 3 (8) | 0 (0) | 0 (0) | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | NA
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | NA
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | NA
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | NA
Dry eye (Eye disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | NA
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Periorbital oedema (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | NA
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Constipation (Gastrointestinal disorders) | 16 (22) | 11 (18) | 0 (0) | 0 (0) | NA
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 2 (3) | 1 (1) | 0 (0) | NA
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Nausea (Gastrointestinal disorders) | 18 (41) | 8 (19) | 1 (1) | 0 (0) | NA
Oral hyperaesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Stomatitis (Gastrointestinal disorders) | 7 (9) | 4 (7) | 0 (0) | 0 (0) | NA
Vomiting (Gastrointestinal disorders) | 2 (4) | 4 (6) | 0 (0) | 0 (0) | NA
Face oedema (General disorders) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | NA
Fatigue (General disorders) | 4 (4) | 5 (7) | 0 (0) | 0 (0) | NA
Infusion site extravasation (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Malaise (General disorders) | 5 (9) | 4 (6) | 0 (0) | 0 (0) | NA
Oedema peripheral (General disorders) | 2 (2) | 5 (6) | 0 (0) | 0 (0) | NA
Puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Pyrexia (General disorders) | 3 (7) | 1 (1) | 1 (1) | 0 (0) | NA
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | NA
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Herpes zoster (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | NA
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | NA
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Nasopharyngitis (Infections and infestations) | 5 (11) | 1 (1) | 0 (0) | 0 (0) | NA
Oral candidiasis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | NA
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | NA
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Alanine aminotransferase increased (Investigations) | 9 (14) | 5 (6) | 0 (0) | 0 (0) | NA
Aspartate aminotransferase increased (Investigations) | 8 (11) | 5 (6) | 0 (0) | 0 (0) | NA
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Blood creatinine increased (Investigations) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | NA
Creatinine renal clearance decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
Lymphocyte count decreased (Investigations) | 7 (22) | 1 (2) | 0 (0) | 0 (0) | NA
Neutrophil count decreased (Investigations) | 7 (14) | 2 (2) | 0 (0) | 0 (0) | NA
Platelet count decreased (Investigations) | 3 (3) | 2 (5) | 0 (0) | 0 (0) | NA
Thyroid hormones decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Thyroxine free increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | NA
Tri-iodothyronine free decreased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | NA
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
White blood cell count decreased (Investigations) | 10 (20) | 3 (4) | 0 (0) | 0 (0) | NA
Decreased appetite (Metabolism and nutrition disorders) | 14 (20) | 9 (23) | 0 (0) | 0 (0) | NA
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | NA
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | NA
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | NA
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
Dysgeusia (Nervous system disorders) | 3 (6) | 5 (9) | 1 (1) | 0 (0) | NA
Headache (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | NA
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | NA
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
Anxiety (Psychiatric disorders) | 1 (2) | 3 (4) | 0 (0) | 0 (0) | NA
Insomnia (Psychiatric disorders) | 6 (8) | 1 (1) | 0 (0) | 0 (0) | NA
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | NA
Hiccups (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 5 (5) | 1 (1) | 0 (0) | NA
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
Alopecia (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
Dry skin (Skin and subcutaneous tissue disorders) | 9 (9) | 2 (2) | 0 (0) | 0 (0) | NA
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | NA
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Hypertension (Vascular disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (2):
  • Study Protocol (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT03950674/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT03950674/SAP_001.pdf